CLINICAL TRIAL: NCT03233243
Title: Rosuvastatin Effect on Atherosclerotic Plaque Metabolism - a Subclinical Atherosclerosis Imaging Study With 18F-NaF PET-CT
Brief Title: Rosuvastatin Effect on Atherosclerotic Plaque Metabolism
Acronym: ROPPET-NAF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Manuel Oliveira Santos, MD, University of Coimbra
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: ICNAS-2016-01
Record Dates: First submitted 2017-07-25; First posted 2017-07-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Molecular Imaging
Keywords: Rosuvastatin; Sodium fluoride; Positron-emission tomography
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with positive 18F-NaF plaques (Experimental): Patients with 18F-NaF-positive plaques (coronary, aortic or carotid) with TBR > 1.5
  Interventions: Drug: Rosuvastatin Oral Tablet
- Patients without 18F-NaF-positive plaques (No Intervention): Subjects without 18F-NaF- positive plaques will be excluded from the pharmacological intervention study

INTERVENTIONS:
Drug: Rosuvastatin Oral Tablet — Patients with 18F-NaF-positive plaques will be treated with 20 mg of rosuvastatin daily for six months, except in patients who need a 55% LDL reduction to achieve recommended targets (rosuvastatin 40 mg). A second visit (visit 2) will take place eight weeks after therapy initiation to monitor for compliance and adverse events report: therapy will be discontinued if there is an elevation of creatine kinase over five times the ULN with myalgia or alanine amino-transferase three times the ULN.
  Arms: Patients with positive 18F-NaF plaques

SUMMARY:
Atherosclerotic plaque uptake of 18F-sodium fluoride (NaF) in positron emission tomography with computed tomography (PET-CT) was recently shown to correlate with clinical instability in patients with CV disease. We hypothesize that rosuvastatin reduces 18F-NaF plaque uptake.

Our group will scan coronary, aortic and carotid arteries of high-risk CV subjects with 18F- NaF-PET-CT. Individuals with 18F-NaF-positive plaques will be treated with rosuvastatin for six months, followed by 18F-NaF-PET-CT re-evaluation.

DETAILED DESCRIPTION:
Background:

Cardiovascular diseases (CVD) are the main cause of mortality in developed countries; its prevention is challenging. Advances in molecular imaging of the atherosclerotic plaque enhanced the study of its pathophysiology, including the positron emission tomography with computed tomography (PET-CT) scan. The marker 18F-sodium fluoride (NaF) has been studied in peripheral arteries plaque imaging as an in vivo marker of on-going calcification. The 18F ions deposit in the bone by exchange of hydroxyl group on the surface of the hydroxyapatite matrix to form fluoroapatite, so this tracer detects areas of active calcification and osteogenic remodeling. Coronary imaging with 18F-NaF labelled PET-CT was recently described and proposed to be able to discriminate between active and inactive coronary calcification, possibly identifying high-risk patients.

Statin therapy is approved for primary and secondary CVD prevention due to both its cholesterol-lowering effect and positive pleiotropic properties in the plaque. In particular, rosuvastatin diminishes mortality and vascular events when used in primary and secondary prevention. High doses of rosuvastatin resulted in atherosclerosis regression as assessed with coronary intravascular ultrasound, carotid intima-media thickness (CIMT) and lipid content reduction of the atherosclerotic plaque (near-infrared spectroscopy analysis).

We do not know the effects of statins in the 18F-NaF uptake.

Design:

Investigator's initiative prospective study of 18F-NaF-PET-CT coronary, aortic and carotid plaques imaging in primary prevention subjects, with a before and after experiment with rosuvastatin treatment and long-term follow-up. The protocol was approved by the Ethics Committee of Faculty of Medicine of the University of Coimbra and written according to Good Clinical Practice and the Declaration of Helsinki.

Taks:

1. Screening - visit 0:

   Patients followed at the Arterial Hypertension clinic of Centro Hospitalar e Universitário de Coimbra will be screened and selected if they meet all of the inclusion criteria.
2. Baseline assessment:

   Clinical questionnaire and standard physical examination. CV risk will be estimated according to SCORE equations and the American Heart Association atherosclerotic cardiovascular disease calculator. Patients' medical history and CV risk factors will be recorded, as well as physical examination findings, including age, race, gender, smoking status (current, past, quantification with pack-years), diabetes mellitus (type 1, 2, pre- diabetes), family history of premature coronary heart disease (first degree: men < 55 and women < 65 years old), relevant past medical history, blood pressure, heart rate, weight and height. Levels of total cholesterol, high and low-density lipoprotein cholesterol (HDL and LDL), triglycerides, creatinine, creatine kinase, alanine amino-transferase, aspartate amino- transferase, gamma-glutamyl transpeptidase, alkaline phosphatase, glycated hemoglobin, fasting glucose, high-sensitivity C-reactive protein and haemoglobin will be determined.
3. Baseline 18F-NaF labelled PET-CT - visit 1:

   Patients will undergo whole body 18F-NaF-PET-CT for identification of coronary, carotid, thoracic and abdominal aorta arteries plaques and quantification of 18F-NaF uptake (tissue-to-background ratio (TBR)). Scans will be reviewed and analysed by experienced observers blinded to the clinical diagnosis. Subjects without 18F-NaF-positive plaques will be excluded from the pharmacological intervention study.
4. Rosuvastatin treatment:

   At visit 1, patients with 18F-NaF-positive plaques will be treated with 20 mg of rosuvastatin daily for six months, except in patients who need a 55% LDL reduction to achieve recommended targets (rosuvastatin 40 mg).
5. Second 18F-NaF labelled PET-CT - visit 3:

Subjects will undergo a second PET-CT scan six months after statin treatment to assess changes in 18F-NaF plaque uptake. Medication compliance will be monitored, as well as adverse events reporting.

Statistical analysis:

18F-NaF uptake after rosuvastatin treatment will be compared to baseline values with paired samples T student test or Wilcoxon text according to the normality of the distribution. Sample size was estimated according to the preliminary results of 25 subjects (pilot study) and the primary endpoint of reducing maximum 18F-NaF uptake as assessed by TBR. Individuals with no significant 18F-NaF uptake were excluded from this analysis (n=4): mean TBR 2.16 and SD 0.40. At 90% power and a significance level of 0.05, assuming a correlation of 0.8 and 10% difference in TBR, the calculated sample size is 32. As only 21 out of 25 subjects in the pilot study displayed criteria for the pharmacological study, it is necessary to perform 44 baseline studies, followed by 36 subjects re-evaluation (drop-out margin of 4 subjects), totaling 80 PET-CT scans.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 40 years;
2. Written informed consent;
3. Considered to be at high or very high CV risk according to the European Society of Cardiology guidelines, fulfilling any of the following criteria:

   * predicted fatal CV event at 10 years ≥5% (SCORE tables for low-risk countries);
   * chronic kidney disease with glomerular filtration rate (GFR) under 60 mL/min (Modification of Diet in Renal Disease equation - MDRD);
   * diabetes mellitus (type 1 or 2);
   * markedly elevated single risk factors.

Exclusion Criteria:

* Previous CV events;
* GFR under 30 mL/min;
* Known hepatic dysfunction or alanine amino-transferase level more than twice the upper limit of the normal (ULN) range;
* Creatine kinase level more than three times the ULN;
* Known myopathy;
* Statin hypersensivity;
* Hormone replacement therapy;
* Malignant neoplasms in the past five years (excluding basal-cell skin carcinoma);
* Uncontrolled hypothyroidism;
* Chronic inflammatory disease (such as rheumatoid arthritis, inflammatory bowel disease);
* Pregnancy or women in child bearing age without contraceptive;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Variation in 18F-NaF uptake in coronary, aortic and carotid plaques (tissue to background ratio - TBR) | 6 months
  * Whole body 18F-NaF-PET-CT for identification of coronary, carotid, thoracic and abdominal aorta arteries plaques:
  * administration of 125 MBq 18F-NaF intravenously, followed by an attenuation correction CT scan and PET imaging after 60 min. Coronary images will be reconstructed according with the usual protocol of PET-CT. Two-dimensional regions of interest will be drawn around all major epicardial coronary vessels and around the major vessels on three millimetres axial slices.
  * Quantification of 18F-NaF uptake at baseline and after optimal treatment including statins:
  * ratio of the maximum standard uptake value (SUV) in the region of interest (the decay corrected tissue concentration of the tracer divided by the injected dose per bodyweight) and blood pool activity in the superior vena cava: tissue-to-background ratio (TBR).
  * Primary outcome: variation in maximum TBR at any vascular territory (coronary, carotid or aortic)

SECONDARY OUTCOMES:
Variation in 18F-NaF uptake in coronary, aortic and carotid plaques (corrected uptake per lesion - CUL) | 6 months
  * Quantification of 18F-NaF uptake at baseline and after optimal medical treatment
  * difference between the maximum SUV in the region of interest and blood pool activity in the superior vena cava: corrected uptake per lesion - CUL.
  * Primary outcome: variation in maximum CUL at any vascular territory (coronary, carotid or aorta)

OTHER OUTCOMES:
Safety outcome | 6 months
  Adverse events monitoring related with medical treatment namely statins: myalgia, myopathy (CK), hepatotoxicity (ALT), gastrointestinal symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Castelo-Branco, PhD, Study Director — Coimbra's University - Faculty of Medicine
Locations (1):
- Centro Hospitalar e Universitário de Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dweck MR, Chow MW, Joshi NV, Williams MC, Jones C, Fletcher AM, Richardson H, White A, McKillop G, van Beek EJ, Boon NA, Rudd JH, Newby DE. Coronary arterial 18F-sodium fluoride uptake: a novel marker of plaque biology. J Am Coll Cardiol. 2012 Apr 24;59(17):1539-48. doi: 10.1016/j.jacc.2011.12.037. PMID 22516444
- [Background] Joshi NV, Vesey AT, Williams MC, Shah AS, Calvert PA, Craighead FH, Yeoh SE, Wallace W, Salter D, Fletcher AM, van Beek EJ, Flapan AD, Uren NG, Behan MW, Cruden NL, Mills NL, Fox KA, Rudd JH, Dweck MR, Newby DE. 18F-fluoride positron emission tomography for identification of ruptured and high-risk coronary atherosclerotic plaques: a prospective clinical trial. Lancet. 2014 Feb 22;383(9918):705-13. doi: 10.1016/S0140-6736(13)61754-7. Epub 2013 Nov 11. PMID 24224999
- [Background] Blomberg BA, Thomassen A, de Jong PA, Simonsen JA, Lam MG, Nielsen AL, Mickley H, Mali WP, Alavi A, Hoilund-Carlsen PF. Impact of Personal Characteristics and Technical Factors on Quantification of Sodium 18F-Fluoride Uptake in Human Arteries: Prospective Evaluation of Healthy Subjects. J Nucl Med. 2015 Oct;56(10):1534-40. doi: 10.2967/jnumed.115.159798. Epub 2015 Jul 23. PMID 26205304
- [Background] Oliveira-Santos M, Castelo-Branco M, Silva R, Gomes A, Chichorro N, Abrunhosa A, Donato P, Pedroso de Lima J, Pego M, Goncalves L, Ferreira MJ. Atherosclerotic plaque metabolism in high cardiovascular risk subjects - A subclinical atherosclerosis imaging study with 18F-NaF PET-CT. Atherosclerosis. 2017 May;260:41-46. doi: 10.1016/j.atherosclerosis.2017.03.014. Epub 2017 Mar 10. PMID 28349887
- [Background] Ferreira MJV, Oliveira-Santos M, Silva R, Gomes A, Ferreira N, Abrunhosa A, Lima J, Pego M, Goncalves L, Castelo-Branco M. Assessment of atherosclerotic plaque calcification using F18-NaF PET-CT. J Nucl Cardiol. 2018 Oct;25(5):1733-1741. doi: 10.1007/s12350-016-0776-9. Epub 2017 Jan 9. PMID 28070735